CLINICAL TRIAL: NCT06836414
Title: Early Cancer Detection in Firefighters With Low-Dose Chest CT: A Community-Based Approach
Brief Title: Lung Cancer Screening CT for Firefighters
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Hayward Firefighters Local 1909 of the International Association of Firefighters (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24053; NCI-2025-00336 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2025-02-14; First posted 2025-02-20 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Smoke Inhalation; Exposure, Inhalation; Exposure to Pollution; Exposure Occupational; Lung Diseases; Lung Cancer; Lung Diseases, Interstitial; Occupational Exposure; Occupational Lung Disease; Interstitial Lung Disease
Keywords: Population research; Cancer Screening
MeSH Terms: conditions — Smoke Inhalation Injury; Respiratory Aspiration; Lung Diseases; Lung Neoplasms; Lung Diseases, Interstitial | interventions — Surveys and Questionnaires; Health Records, Personal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Firefighters (Lung Screening CT) (Other): Participants will receive a single, low-dose, chest CT without contrast as indicated for lung cancer screening. Participants will be followed up for at least 1 year following the scan and have ongoing medical record reviews.
  Interventions: Procedure: Low-dose Computerized tomography (CT) of Chest; Other: Questionnaires; Other: Medical History
- Firefighters with Previously Diagnosed Malignancy (Other): Participants with a history of cancer will have a medical record review as part of a case-control cohort.
  Interventions: Other: Medical History

INTERVENTIONS:
Procedure: Low-dose Computerized tomography (CT) of Chest — Undergo CT for lung cancer screening
  Other Names: Chest CT; Chest CT Scan; Low-dose Chest CT
  Arms: Firefighters (Lung Screening CT)
Other: Questionnaires — Participants will complete questionnaires on or before the day of the scan.
  Arms: Firefighters (Lung Screening CT)
Other: Medical History — Medical history will be obtained in person and via medical record review
  Other Names: Medical Record Review; Medical Chart Review

SUMMARY:
Firefighters are at increased risk for cancer due to exposure to carcinogenic substances. Current lung cancer screening guidelines are predominantly based on smoking history and do not take into account high risk occupational exposures such as firefighting. This study aims to provide chest computed tomography (CT) scans to firefighters to determine the prevalence of lung cancer, other cancers detectable on CT chest, and lung diseases associated with increased cancer risk.

DETAILED DESCRIPTION:
This is a single-group prospective interventional study and a community-based participatory project led by University of California, San Francisco and in close collaboration with the firefighter community in California.

PRIMARY OBJECTIVE:

I. Determine the prevalence of lung cancer, other cancers and cancer risk factors detectable on chest Computerized Tomography (CT) (Aim 1).

II. Identify imaging and non-imaging predictors of lung cancer and other cancers detectable on chest CT.

SECONDARY OBJECTIVE:

I. Determine the prevalence of incidental findings on chest CT (Aim 1).

II. Determine the risk factors for cancer development in firefighters (Aim 2).

EXPLORATORY OBJECTIVES:

I. Long term follow-up to determine the incidence of lung cancer and other cancers among firefighters.

II. Develop a firefighter cancer imaging registry.

OUTLINE:

Participants will be administered a single, low dose chest CT to included participants and collect comprehensive demographic, clinical, and occupational data. Participants will be followed up at 1-2 months, for at least 1 year and up to 10 years to collect any follow-up imaging and biopsy results, if applicable.

ELIGIBILITY:
Inclusion Criteria:

1. Age 35 years or greater. If the participant is above the age of 80, participants must be otherwise healthy and well-fit to undergo treatment if lung cancer were to be discovered.
2. Never smoker or quit more than 15 years ago.
3. Able to understand study procedures and to comply with them for the entire length of the study.
4. Ability of individual or legal guardian/representative to understand a written informed consent document, and the willingness to sign it.
5. Length in profession for 10 or more years. This includes both volunteer firefighting and professional firefighting, self-attested as verifiable by professional records.

Additional cases for Aim 2:

1. Age 18+, may include deceased firefighters.
2. A previous or current history of confirmed thoracic malignancy (except localized skin cancer, cancer in situ, or other localized cancers)

Exclusion Criteria:

* Aim 1:

  1. Contraindication to any study-related procedure or assessment.
  2. Personal history of malignancy within 5 years (except localized skin cancer, cancer in situ, or localized cancers that are definitively treated and are unlikely to recur) or lung cancer at any time.
  3. Participants will be assessed for active pregnancy per standard procedure for clinical lung cancer screening CT at University of California, San Francisco which includes asking the participants directly along with documentation of whether the negative pregnancy was self-reported or confirmed with a urine pregnancy test.
  4. Prior CT chest within 1 year.
  5. Symptoms highly suggestive of lung cancer, including unexplained weight loss of over 30 pounds (lbs) within the past 12 months or unexplained hemoptysis.
* Aim 2:

No exclusion criteria

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with detected lung cancers (Aim 1) | Up to 10 years
  The proportion of participants with detected lung cancers will be determined by the frequency of image findings that indicate lung cancer, and an ultimate clinical diagnosis associated with the imaging finding.
Proportion of participants with detected other cancers (Aim 1) | Up to 10 years
  The proportion of participants with detected cancers, other than lung, will be determined by the frequency of image findings that indicate other cancer, and an ultimate clinical diagnosis associated with the imaging finding.
Proportion of participants with occupational lung disease (Aim 1) | Up to 10 years
  Occupational or work-related lung diseases are lung conditions that have been caused or made worse by long-term exposure to certain irritants in the workplace. The proportion of participants with occupational lung disease will be determined by the frequency of image findings that indicate occupationally associated lung disease, and an ultimate clinical diagnosis associated with the imaging finding.
Proportion of participants with diagnosed interstitial lung disease (Aim 1) | Up to 10 years
  Interstitial Lung Disease (ILD) is a group of diseases that irritate, inflame, or scar the lungs and supporting air sacs. The proportion of participants with diagnosed interstitial lung disease will be determined by the frequency of image findings that indicate ILD, and an ultimate clinical diagnosis associated with the imaging finding.
Number of participants within of each Lung-RADS risk group | Up to 10 years
  The Lung CT Screening Reporting and Data System (Lung-RADS) is a measure developed by the American College of Radiologists to standardize the reporting and management of screen-detected pulmonary nodules. Nodules are categorized as 0=Incomplete, 1=Negative, 2=Benign Appearance or Behavior, 3=Probably Benign, or 4A /4B /4X = Suspicious with an additional modifier of S=Other or C=Prior Lung Cancer to be added to the 4 category codes as needed. The frequency of participants within each Lung-RADS risk group as determined by imaging procedures will be reported.

SECONDARY OUTCOMES:
Percentage of participants with incidental clinical findings | Up to 10 years
  The percentage of participants with incidental findings be determined by the frequency of image findings that indicate presence of possible coronary calcium, aortic aneurysm, thyroid nodules, liver pathology and osseous pathology and an ultimate clinical diagnosis associated with the imaging finding.
Number of risk factors identified as associated with cancer development | Up to 10 years
  The number of not-yet identified risk factors that are determined to be significantly associated with the development of thoracic cancers will be determined using logistic regression methods.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Ho Sohn, MD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No